CLINICAL TRIAL: NCT02468713
Title: An Open Label, Randomized, Single Dose, Crossover Study to Evaluate the Effect on Blood Lipid Profiles of Omega-3 Enriched Total Parenteral Nutrition in Healthy Korean Male Subjects
Brief Title: Effect on Blood Chemistry and Inflammatory Marker of Omega-3 Enriched Total Parenteral Nutrition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Hee Chul Yu, Professor, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CUH201412002
Record Dates: First submitted 2015-05-29; First posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Omega-3; Blood lipid profiles; DHA; EPA; Triglyceride; Glucose; Insulin; LDL; TPN
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Combiflex® lipid peri as a reference product (Period 1) -> Winuf® peri as a test product (Period 2)
  Interventions: Drug: Combiflex® lipid peri; Drug: Winuf® peri
- Group 2 (Experimental): Winuf® peri as a test product (Period 1) -> Combiflex® lipid peri as a reference product (Period 2)
  Interventions: Drug: Combiflex® lipid peri; Drug: Winuf® peri

INTERVENTIONS:
Drug: Combiflex® lipid peri — total parenteral nutrition solutions containing glucose, amino acids, electrolyte, soybean oil
Drug: Winuf® peri — total parenteral nutrition solution containing glucose, amino acids, electrolyte, soybean oil, medium chain triglyceride, olive oil and fish oil

SUMMARY:
Fish oil is a rich source of omega-3 fatty acids, especially eicosapentanoic acid and docosahexaenoic acid, and it is not used widely in parenteral nutrition because fish oil emulsions have not been commercially available until very recently. The Objective of this study is to to evaluate the effect on blood lipid profiles of omega-3 enriched total parenteral nutrition in healthy Korean male subjects. This study is designed as a randomized, open-label, 2-treatment, 2-way crossover trial. Blood samples will be collected every 1 hour from 0 to 12 hours after starting an intravenous infusion for triglyceride, glucose, and insulin.

DETAILED DESCRIPTION:
Fish oil is a rich source of omega-3 fatty acids, especially eicosapentanoic acid and docosahexaenoic acid, and it is not used widely in parenteral nutrition because fish oil emulsions have not been commercially available until very recently. The Objective of this study is to to evaluate the effect on blood lipid profiles of omega-3 enriched total parenteral nutrition in healthy Korean male subjects.

This study is designed as a randomized, open-label, 2-treatment, 2-way crossover trial. The 16 subjects will be randomly assigned to 1 of 2 sequences of the two treatments: Combiflex® lipid peri or Winuf® peri will be infused via peripheral venous catheter for 6 hours at 3 ml/kg/h. Blood samples will be collected every 1 hour from 0 to 12 hours after starting an intravenous infusion for triglyceride, glucose, and insulin. Cholesterol, HDL-cholesterol, LDL-cholesterol, AST, ALT, and total bilirubin as liver function biomarkers, and hsCRP as inflammatory biomarker will be analysed at 0, 6 and 12 hour after starting an intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 30 and 55 years
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg
* An informed consent document signed and dated by the subject
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Screening sitting blood pressure >150 mm Hg (systolic) or >90 mm Hg (diastolic)
* Use of tobacco in excess of the equivalent of 20 cigarettes per day
* Use of prescription or nonprescription drugs within 10 days
* Blood donation within 2 months prior to dosing, or plasma donation within 1 month prior to dosing
* Severe hyperlipidemic patients
* Severe liver failure patients

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To compare AUC of plasma triglyceride between Winuf peri and Combiflex lipid peri | Before-dosing(0 hour) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing
  The wash-out period will be 7 days, and the second study period will be conducted on the same schedule as the first study period, with the exception of the assignment of the investigational product.
To compare Cmax of plasma triglyceride between Winuf peri and Combiflex lipid peri | Before-dosing(0 hour) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing
  The wash-out period will be 7 days, and the second study period will be conducted on the same schedule as the first study period, with the exception of the assignment of the investigational product.

SECONDARY OUTCOMES:
To compare AUC of plasma glucose between Winuf peri and Combiflex lipid peri | Before-dosing(0 hour) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing
To compare Cmax of plasma glucose between Winuf peri and Combiflex lipid peri | Before-dosing(0 hour) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing
To compare AUC of plasma insulin between Winuf peri and Combiflex lipid peri | Before-dosing(0 hour) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing
To compare Cmax of plasma insulin between Winuf peri and Combiflex lipid peri | Before-dosing(0 hour) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing
To compare AUC of plasma omega-3 between Winuf peri and Combiflex lipid peri | Before-dosing(0 hour) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing
To compare Cmax of plasma omega-3 between Winuf peri and Combiflex lipid peri | Before-dosing(0 hour) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours after dosing
Change from baseline in blood cholesterol level at 6 and 12 hours | Before-dosing(0 hour) and 6, and 12 hours
Change from baseline in blood HDL-cholesterol level at 6 and 12 hours | Before-dosing(0 hour) and 6, and 12 hours
Change from baseline in blood LDL-cholesterol level at 6 and 12 hours | Before-dosing(0 hour) and 6, and 12 hours
Change from baseline in blood AST level at 6 and 12 hours | Before-dosing(0 hour) and 6, and 12 hours
Change from baseline in blood ALT level at 6 and 12 hours | Before-dosing(0 hour) and 6, and 12 hours
Change from baseline in blood total bilirubin level at 6 and 12 hours | Before-dosing(0 hour) and 6, and 12 hours
Change from baseline in blood hsCRP level at 6 and 12 hours | Before-dosing(0 hour) and 6, and 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hee Chul Yu, MD, PhD, Principal Investigator — Professor
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea